CLINICAL TRIAL: NCT01011621
Title: Comparative Evaluation of the Efficacy and Tolerability of Prednisolone Acetate 0.5% Cream Versus Betamethasone Valerate 0.1% Cream in the Treatment of Pediatric and Adult Dermatosis
Brief Title: Efficacy and Tolerability of Prednisolone Acetate 0.5% Cream Versus Betamethasone Valerate 0.1% Cream in Cortisosensitive Dermatosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mantecorp Industria Quimica e Farmaceutica Ltd. (Industry)
Responsible Party: Celso Pereira Sustovich, Medical Director, Mantecorp Indústria Química e Farmacêutica Ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE/P/08-1
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2009-11-11 (Estimated); Status verified 2009-11

CONDITIONS: Dermatitis, Atopic; Dermatitis, Contact; Dermatitis, Seborrheic; Psoriasis
Keywords: Prednisolone acetate; Betamethasone valerate
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis, Contact; Dermatitis, Seborrheic; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 0.5% prednisolone acetate cream (Experimental)
  Interventions: Drug: 0.5% prednisolone acetate cream
- 0.1% betamethasone valerate cream (Active Comparator)
  Interventions: Drug: 0.1% betamethasone valerate cream

INTERVENTIONS:
Drug: 0.5% prednisolone acetate cream — Small amount applied over the lesion twice a day for 14 days.
  Arms: 0.5% prednisolone acetate cream
Drug: 0.1% betamethasone valerate cream — Small amount applied over the lesion twice a day for 14 days.
  Arms: 0.1% betamethasone valerate cream

SUMMARY:
Topical corticosteroids are largely used in dermatology. The major problem related to their use is that the same mechanisms underlying their therapeutic effects (antiinflammatory and antiproliferative) may lead to adverse events. Conditions sensitive to corticosteroids require formulations with mild to moderate potency while high-potency corticosteroids era required in less responsive conditions. The aim of the present study is to compare the safety and efficacy of prednisolone acetate 0.5% cream (mild-potency non-fluoridated corticosteroid) versus betamethasone valerate 0.1% cream (high-potency fluoridated corticosteroid) in the treatment of mild to moderate cortisosensitive dermatosis (atopic dermatitis, contact dermatitis, seborrheic dermatitis and psoriasis). The study hypothesis is that 0.5% prednisolone cream will be as effective as 0.1% betamethasone cream and will be an alternative option to treat corticosensitive dermatosis in body areas where the use of fluoridated corticosteroids is contraindicated, such as the face.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with corticosensitive dermatosis (atopic dermatitis, contact dermatitis, seborrheic dermatitis, psoriasis) mild to moderate in intensity;
* Compliance of the subject to the treatment protocol;
* Agreement with the terms o the informed consent by the participants
* Subjects who did not use the following medicines before inclusion: topical corticosteroids or other therapies to dermatitis (30 days); oral corticosteroids (180 days); parenteral corticosteroids (180 days); immunomodulators/immunosuppressor (30 days); any drug under investigation (1 year); any therapy for the studied clinical conditions (180 days); keratolytic agents (30 days); emollient agents (30 days); tazarotene (30 days); vitamin D (topical or oral, 30 days); methotrexate (30 days); acitretin (2 years); UV light (30 days); PUVA therapy (30 days).

Exclusion criteria:

* Pregnancy or risk of pregnancy
* Lactation
* History of allergy of any component of the formulations
* Other conditions considered by the investigator as reasonable for non-eligibility
* HIV positivity
* Drug abuse
* Subjects without previous response to topical corticosteroids
* Subjects with intense sun exposure within 15 days of the screening

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 170 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate efficacy and safety of 0.5% prednisolone cream in comparison to 0.1% betamethasone cream in the treatment of corticosensitive dermatosis. | 14 days

SECONDARY OUTCOMES:
Evaluate physicians' and patients' perception of the efficacy and tolerability of treatment. | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Mário C Pires, MD, Principal Investigator — Hospital Padre Bento de Guarulhos; Roberta F. J. Criado, MD, Principal Investigator — Faculdade d Medicina do ABC; Adilson Costa, MD, Principal Investigator — KOLderma